CLINICAL TRIAL: NCT02668445
Title: The Effects of Glycogen Availability on the Skeletal Muscle Molecular Response After Concurrent Exercise
Brief Title: Molecular Response After Concurrent Exercise With Low Glycogen
Acronym: Glyconcurrent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL54408.081.15
Record Dates: First submitted 2016-01-26; First posted 2016-01-29 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2016-02

CONDITIONS: Healthy
Keywords: Concurrent; muscle; glycogen; molecular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low carbohydrate (Experimental): Subjects will eat a low carbohydrate diet
  Interventions: Other: Standard meal containing low or high carbohydrate content
- High carbohydrate (Experimental): Subjects will eat a high carbohydrate diet
  Interventions: Other: Standard meal containing low or high carbohydrate content

INTERVENTIONS:
Other: Standard meal containing low or high carbohydrate content

SUMMARY:
This is a randomized, counterbalanced crossover design, in which 14 male subjects will complete two experimental trials. Each trial will be separated by a minimum of at least 12 days (range: 12-30 days). The study aims to investigate the effects of low glycogen availability on skeletal muscle molecular response after a concurrent exercise day.

DETAILED DESCRIPTION:
Two experimental exercise trials; a low carbohydrate (= LOW) and a high carbohydrate (= HIGH) trial. During both experimental days subjects will complete an continues submaximal cycling bout in the morning followed by a resistance exercise session in the early afternoon. During the LOW trial subjects will receive a low carbohydrate mixed meal, during the HIGH trial subjects will be provided with a high carbohydrate meal. In addition, on both experimental days subjects will receive adequate protein beverages. Lastly, protein will be provided post resistance exercise.

ELIGIBILITY:
Inclusion Criteria:

* Male gender between 18 and 30 years of age
* BMI between 18.5 - 25 kg/m2
* Participating in regular exercise training (at least 1 exercise session, and a maximum of 3 exercise session per week)
* Used to different types of exercise (endurance, resistance and/or concurrent)
* Willing to give blood samples
* Willing to give muscle biopsies
* No use of antibiotics during the study or in the past month
* No drug use
* Suitable veins for blood withdrawal
* Registered by a general-practitioner
* Consumption of alcohol beverages is less than 21 per week
* No blood donor during the study
* No vegetarian and willing to eat meat during the experimental days
* Able to be present and participate at both test days and pre testing moments
* Not employed, or intern, or working on thesis at the department of Human Nutrition at Wageningen University
* Not participating in another scientific study (except EetMeetWeet)
* Able to participate during the experimental days en pre tests
* Able to speak Dutch

Exclusion Criteria:

* Medical condition that can interfere with the study outcome (i.e. cardiovascular disease, pulmonary disease, gluten intolerance)
* Systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg
* Use of medications known to interfere with gene expression in the muscles (i.e. statins, fenofibrate)
* Use of antithrombotic therapy (marcoumar, sintromitis).
* Diagnosed diabetes mellitus type 1 or 2
* (Chronic) injuries of the locomotor system that can interfere with the intervention

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Proteins involved in hypertrophy | 10 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Human Nutrition, Wageningen University, Wageningen, Gelderland, Netherlands